CLINICAL TRIAL: NCT01450696
Title: A Randomized, Open Label, Multicenter Phase IIIb Study Comparing Two Trastuzumab Dosing Regimens, Each in Combination With Cisplatin/Capecitabine Chemotherapy, as First-Line Therapy in Patients With HER2-Positive Metastatic Gastric or Gastro-Esophageal Junction Adenocarcinoma Who Have Not Received Prior Treatment for Metastatic Disease
Brief Title: A Study of Herceptin (Trastuzumab) in Combination With Cisplatin/Capecitabine Chemotherapy in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Metastatic Gastric or Gastro-Esophageal Junction Cancer
Acronym: HELOISE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: futility following planned interim analysis
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO27798; 2011-001526-19 (EudraCT Number)
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin; Trastuzumab

ARMS (2):
- Capecitabine + Cisplatin + Herceptin (6 mg/kg) (Active Comparator): Participants will receive Herceptin at a loading dose of 8 mg/kg on Day 1 of Cycle 1 followed by 6 mg/kg q3w as a standard of care from Day 1 of Cycle 2 until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason (cycle length = 21 days). Participants will also receive cisplatin 80 mg/m^2 intravenously q3w plus capecitabine 800 mg/m^2 orally twice daily for 14 days q3w for up to 6 treatment cycles (Cycles 1 to 6).
  Interventions: Drug: Capecitabine; Drug: Cisplatin; Drug: Herceptin
- Capecitabine + Cisplatin + Herceptin (10 mg/kg) (Experimental): Participants will receive Herceptin at a loading dose of 8 mg/kg on Day 1 of Cycle 1 followed by 10 mg/kg q3w from Day 1 of Cycle 2 until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason (cycle length = 21 days). Participants will also receive cisplatin 80 mg/m^2 intravenously q3w plus capecitabine 800 mg/m^2 orally twice daily for 14 days q3w for up to 6 treatment cycles (Cycles 1 to 6).
  Interventions: Drug: Capecitabine; Drug: Cisplatin; Drug: Herceptin

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be administered at a dose of 800 mg/m^2 orally twice daily for 14 days q3w for up to 6 cycles (Cycles 1 to 6).
Drug: Cisplatin — Cisplatin will be administered at a dose of 80 mg/m^2 intravenously q3w on Day 1 of each 3-week cycle for up to 6 cycles (Cycles 1 to 6).
Drug: Herceptin — Herceptin will be administered at a loading dose of 8 mg/kg on Day 1 of Cycle 1 followed by 6 or 10 mg/kg (depending upon treatment assignment) q3w from Day 1 of Cycle 2 until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason.
  Other Names: Trastuzumab

SUMMARY:
This randomized, open-label, multicenter, international Phase IIIb study will compare the efficacy and safety of two Herceptin dosing regimens in combination with cisplatin/capecitabine chemotherapy in participants with HER2-positive metastatic gastric or gastro-esophageal junction adenocarcinoma. Participants who have not received prior treatment for metastatic disease will be randomized to receive Herceptin intravenously as either an 8-milligram per kilogram (mg/kg) loading dose followed by 6 mg/kg every 3 weeks (q3w) as standard of care or an 8-mg/kg loading dose followed by 10 mg/kg q3w until disease progression. Capecitabine will be administered for 6 cycles at a dose of 800 milligrams per meter-squared (mg/m^2) orally twice a day on Days 1 to 14 of each 3-week cycle, and cisplatin will be administered intravenously for 6 cycles at a dose of 80 mg/m^2 on Day 1 of each 3-week cycle. Herceptin will be continued until disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the stomach or gastro-esophageal junction with metastatic disease documented to involve at least liver or lung or both
* Measurable disease according to RECIST Version 1.1 or non-measurable evaluable disease
* At least 2 organs involved in metastatic gastric tumor (including at least lung or liver or both) in addition to the site of primary tumor, where metastasis in distant lymph nodes, peritoneal metastasis, and malignant pleural effusion may count as "organs" in this context
* HER2-positive primary or metastatic tumor as assessed by central laboratory
* Adequate renal function (creatinine clearance greater than equal to (≥) 45 milliliters per minute [mL/min])
* Eastern Cooperative Oncology Group (ECOG) performance status of 2

Exclusion Criteria:

* Previous chemotherapy for locally advanced or metastatic disease
* Prior gastrectomy (partial or total) for the underlying malignant disease under investigation
* Prior therapy with an anti-HER2 agent and/or platinum-based chemotherapeutic agent
* Residual relevant toxicity resulting from previous therapy
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome (such as jejunostomy probe and gastric or jejunostomy tubes) which may impair the ability to administer or absorb capecitabine
* Current (significant or uncontrolled) gastrointestinal bleeding
* Other malignancy within the last 5 years, except for carcinoma in situ of the cervix and basal or squamous cell carcinoma of the skin
* History of documented congestive heart failure, angina pectoris requiring medication, electrocardiogram (ECG) evidence of transmural myocardial infraction, poorly controlled hypertension, clinically significant valvular heart disease, or high-risk uncontrollable arrhythmias
* Baseline left ventricular ejection fraction (LVEF) less than (<) 50%, documented by echocardiography, multiple-gated radionuclide angiography (MUGA) scan, or cardiac magnetic resonance imaging (MRI)
* Chronic or high-dose corticosteroid therapy
* History or clinical evidence of brain metastases
* Pregnant women
* Active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C, or HIV-seropositive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (100):
- United States (8):
  - La Jolla, California
  - Los Angeles, California
  - Whittier, California
  - Goshen, Indiana
  - Wichita, Kansas
  - New York, New York
  - Portland, Oregon
  - Charleston, South Carolina
- Australia (4):
  - Port Macquarie, New South Wales
  - Wahroonga, New South Wales
  - Woodville South, South Australia
  - Murdoch, Western Australia
- Bosnia and Herzegovina (2):
  - Banja Luka
  - Sarajevo
- Brazil (5):
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Barretos, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
- Chile (2):
  - Santiago
  - Viña del Mar
- China (10):
  - Beijing
  - Changchun
  - Changsha
  - Changzhou
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Wuhan
  - Zhengzhou
- Czechia (3):
  - Brno
  - Olomouc
  - Prague
- Germany (3):
  - Berlin
  - Frankfurt
  - Mannheim
- Hungary (5):
  - Budapest
  - Pécs
  - Szolnok
  - Szombathely
  - Veszprém
- Italy (9):
  - Catanzaro, Calabria
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Milan, Lombardy
  - Ancona, The Marches
  - Florence, Tuscany
  - Pisa, Tuscany
- Mexico (4):
  - Distrito Federal
  - Mexico City
  - Monterrey
  - Oaxaca City
- Auckland, New Zealand
- Panama City, Panama
- Peru (3):
  - Arequipa
  - Lima
  - Trujillo
- Philippines (2):
  - Manila
  - Pasig
- Poland (4):
  - Krakow
  - Lublin
  - Warsaw
  - Wieliszew
- Porto, Portugal
- Russia (6):
  - Ivanovo
  - Omsk
  - Ryazan
  - Saint Petersburg
  - Stavropol
  - Tula
- Serbia (3):
  - Belgrade
  - Kamenitz
  - Niš
- South Africa (3):
  - Bloemfontein
  - Cape Town
  - Johannesburg
- South Korea (3):
  - Bundang City
  - Incheon
  - Seoul
- Spain (2):
  - Barcelona, Barcelona
  - Madrid, Madrid
- Turkey (Türkiye) (6):
  - Adana
  - Gaziantep
  - Istanbul
  - Izmir
  - Malatya
  - Sıhhiye, Ankara
- Ukraine (6):
  - Cherkassy
  - Chernivtsi
  - Dnipropetrovsk
  - Donetsk
  - Kiev
  - Lviv
- United Kingdom (4):
  - Denbighshire
  - Leicester
  - Southampton
  - Wolverhampton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 248 participants (124 participants per arm) were randomized in the study up to data cutoff date of 13 February 2015, and 48 additional participants (24 participants per arm) were randomized between data cutoff date of 13 February 2015 and end of study (25 August 2015) for additional safety data.
Groups:
- Capecitabine + Cisplatin + Herceptin (6 mg/kg): Participants received Herceptin at a loading dose of 8 milligrams per kilogram (mg/kg) on Day 1 of Cycle 1 followed by 6 mg/kg every three weeks (q3w) as standard of care from Day 1 of Cycle 2 until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason (cycle length = 21 days). Participants also received cisplatin 80 milligrams per meter-squared (mg/m^2) intravenously q3w plus capecitabine 800 mg/m^2 orally twice daily for 14 days q3w for up to 6 treatment cycles (Cycles 1 to 6).
- Capecitabine + Cisplatin + Herceptin (10 mg/kg): Participants received Herceptin at a loading dose of 8 mg/kg on Day 1 of Cycle 1 followed by 10 mg/kg q3w from Day 1 of Cycle 2 until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason (cycle length = 21 days). Participants also received cisplatin 80 mg/m^2 intravenously q3w plus capecitabine 800 mg/m^2 orally twice daily for 14 days q3w for up to 6 treatment cycles (Cycles 1 to 6).
Period: Overall Study
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Started | 148 | 148
Treated (Safety Population) | 147 | 147
Completed | 0 | 0
Not Completed | 148 | 148
Not completed — Never Treated | 1 | 1
Not completed — Death | 77 | 84
Not completed — Lost to Follow-up | 3 | 3
Not completed — Non-Compliance | 1 | 0
Not completed — Withdrawal by Subject | 13 | 2
Not completed — Study Terminated by Sponsor | 53 | 58

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) population included all participants who were randomized in this study.
Groups:
- Capecitabine + Cisplatin + Herceptin (6 mg/kg): Participants received Herceptin at a loading dose of 8 mg/kg on Day 1 of Cycle 1 followed by 6 mg/kg q3w as standard of care from Day 1 of Cycle 2 until disease progression, occurrence of unacceptable toxicity, or withdrawal from the study for another reason (cycle length = 21 days). Participants also received cisplatin 80 mg/m^2 intravenously q3w plus capecitabine 800 mg/m^2 orally twice daily for 14 days q3w for up to 6 treatment cycles (Cycles 1 to 6).
- Total: Total of all reporting groups
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg) | Total
Number analyzed (Participants) | 148 | 148 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (10.6) | 62.4 (10.7) | 60.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 69
  Male | 116 | 111 | 227

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died - FAS
Description: The percentage of participants who died as of the analysis data cutoff date of 13 February 2015 was reported among participants from the FAS with available data.
Time Frame: From date of randomization until death or premature withdrawal (up to approximately 31 months or data cutoff date of 13 February 2015)
Population: FAS population. Here, number of participants analyzed reflects the number of participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 124 | 124
percentage of participants | 46.8 | 54.0

2. Primary Outcome: Overall Survival - FAS
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause. Overall survival was estimated among participants from the FAS using the Kaplan-Meier approach. The 95 percent (%) confidence interval (CI) for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 124 | 124
months | 12.485 [10.086 to 13.864] | 10.612 [9.363 to 12.419]
Statistical Analysis 1: Comparison: Capecitabine + Cisplatin + Herceptin (6 mg/kg) vs Capecitabine + Cisplatin + Herceptin (10 mg/kg); Stratified analysis included stratum of creatinine clearance (45 to 59 milliliters per minute [mL/min] and greater than or equal to [≥] 60 mL/min). Hazard ratio was estimated by Cox regression; Test type: Superiority or Other; p = 0.2401, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.86 to 1.78]
Statistical Analysis 2: Comparison: Capecitabine + Cisplatin + Herceptin (6 mg/kg) vs Capecitabine + Cisplatin + Herceptin (10 mg/kg); Unstratified analysis. Hazard ratio was estimated by Cox regression; Test type: Superiority or Other; p = 0.1285, Log Rank; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.92 to 1.88]

3. Secondary Outcome: Percentage of Participants Who Died - Per Protocol Set (PPS)
Description: The percentage of participants who died as of the analysis data cutoff date of 13 February 2015 was reported among participants from the PPS.
Time Frame: as for outcome 1
Population: The PPS included all participants who were found to have a trastuzumab minimum plasma concentration (Cmin) less than (<) 12 micrograms per milliliter (μg/mL) on treatment Day 21 of Cycle 1 following the initial loading dose of 8 mg/kg.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 33 | 32
percentage of participants | 51.5 | 59.4

4. Secondary Outcome: Overall Survival - PPS
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause. Overall survival was estimated among participants from the PPS using the Kaplan-Meier approach. The 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 1
Population: PPS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 33 | 32
months | 10.809 [8.082 to 14.752] | 9.363 [5.552 to 14.357]
Statistical Analysis 1: Comparison: Capecitabine + Cisplatin + Herceptin (6 mg/kg) vs Capecitabine + Cisplatin + Herceptin (10 mg/kg); Stratified analysis included stratum of creatinine clearance (45 to 59 mL/min and ≥60 mL/min). Hazard ratio was estimated by Cox regression; Test type: Superiority or Other; p = 0.9931, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.49 to 2.04]
Statistical Analysis 2: Comparison: Capecitabine + Cisplatin + Herceptin (6 mg/kg) vs Capecitabine + Cisplatin + Herceptin (10 mg/kg); Unstratified analysis. Hazard ratio was estimated by Cox regression; Test type: Superiority or Other; p = 0.9458, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.52 to 2.02]

5. Secondary Outcome: Percentage of Participants With Disease Progression or Death - PPS
Description: Disease progression was defined by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as a ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including Baseline (nadir). In addition to the relative increase of 20%, the sum was also required to demonstrate an absolute increase of ≥5 millimeters (mm). The percentage of participants who died or experienced disease progression as of the analysis data cutoff date of 13 February 2015 was reported among participants from the PPS.
Time Frame: From date of randomization until first occurrence of disease progression or death; assessed every 6 weeks (up to approximately 31 months or data cutoff date of 13 February 2015)
Population: PPS population.
Measure: Number; unit: percentage of participants
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 33 | 32
percentage of participants | 75.8 | 81.3

6. Secondary Outcome: Progression-Free Survival - PPS
Description: Progression-free survival was defined as the time between the day of randomization and the date of first documentation of disease progression or date of death, whichever occurred first, measured following RECIST Version 1.1 criteria. Disease progression was defined as a ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including Baseline (nadir). In addition to the relative increase of 20%, the sum was also required to demonstrate an absolute increase of ≥5 mm. The 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: as for outcome 5
Population: PPS population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 33 | 32
months | 5.388 [2.793 to 7.721] | 4.370 [2.727 to 6.834]
Statistical Analysis 1: Comparison: Capecitabine + Cisplatin + Herceptin (6 mg/kg) vs Capecitabine + Cisplatin + Herceptin (10 mg/kg); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.6759, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.63 to 2.02]
Statistical Analysis 2: Comparison: Capecitabine + Cisplatin + Herceptin (6 mg/kg) vs Capecitabine + Cisplatin + Herceptin (10 mg/kg); Unstratified analysis. Hazard ratio was estimated by Cox regression; Test type: Superiority or Other; p = 0.5764, Log Rank; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.67 to 2.05]

7. Secondary Outcome: Percentage of Participants With Objective Response - PPS
Description: Objective response was defined as the occurrence of either a complete response (CR) or partial response (PR) as determined by RECIST Version 1.1 based on investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) were required to have reduction in short axis to <10 mm. PR was defined as a ≥30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters. The 95% CI was constructed using Blyth-Still-Casella method.
Time Frame: as for outcome 5
Population: PPS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 33 | 32
percentage of participants | 57.6 [40.12 to 73.16] | 50.0 [31.89 to 68.11]
Statistical Analysis 1: Comparison: Capecitabine + Cisplatin + Herceptin (6 mg/kg) vs Capecitabine + Cisplatin + Herceptin (10 mg/kg); The 95% CI for difference in response rates was constructed using the normal approximation to the binomial distribution; Test type: Superiority or Other; p = 0.5402, Chi-squared; Difference in response rates = -7.58, 95% CI 2-sided [-31.75 to 16.60]
Statistical Analysis 2: Comparison: Capecitabine + Cisplatin + Herceptin (6 mg/kg) vs Capecitabine + Cisplatin + Herceptin (10 mg/kg); Test type: Superiority or Other; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.28 to 1.96]

8. Secondary Outcome: Trastuzumab Cmin on Day 21 of Cycles 1 to 11 - FAS
Description: Cmin samples were obtained in all participants randomized to receive Herceptin (FAS). The observed Cmin was recorded, averaged among all participants, and expressed in μg/mL.
Time Frame: Day 21 of Cycle 1, 2, 3, 4, 5, 7, 9, 11 (cycle length = 21 days)
Population: FAS population. Here, number of participants analyzed reflects the number of participants who were evaluable for this outcome measure. Here also, "n" reflects the number of participants who were evaluable for each category in the respective arms.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 100 | 99
μg/mL
  Cycle 1 (n=100,99) | 17.1 (14.3) | 18.1 (18.1)
  Cycle 2 (n=93,76) | 19.2 (8.8) | 35.3 (19.4)
  Cycle 3 (n=77,71) | 23.2 (11.8) | 40.7 (20.6)
  Cycle 4 (n=73,61) | 25.9 (12.1) | 47.6 (20.2)
  Cycle 5 (n=70,60) | 26.7 (10.6) | 49.3 (23.2)
  Cycle 7 (n=51,44) | 31.4 (14.2) | 58.1 (27.6)
  Cycle 9 (n=31,24) | 33.7 (17.6) | 61.0 (23.9)
  Cycle 11 (n=24,16) | 32.5 (14.7) | 68.4 (35.9)

9. Secondary Outcome: Trastuzumab Serum Concentration on Day 1 of Cycle 1 - FAS
Description: Trastuzumab serum concentration samples were obtained in all participants randomized to receive Herceptin (FAS). The observed concentration values were recorded, averaged among all participants, and expressed in μg/mL.
Time Frame: Pre-dose (0 minutes) and within 15 minutes after end of 2-hour Herceptin infusion on Day 1 of Cycle 1 (cycle length = 21 days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Number analyzed (Participants) | 110 | 111
μg/mL
  Pre-dose (n=109,110) | 0.168 (1.69) | 0.0204 (0.123)
  End of infusion (n=110,111) | 126 (59.6) | 137 (55.7)

ADVERSE EVENTS:
Time Frame: From date of randomization until 6 months after last dose of study drug or end of study (up to approximately 32 months or final data collection date of 25 August 2015)
Description: Safety evaluable population included all participants who were randomized and received at least one dose of any component of study treatment.
Arm/Group | Capecitabine + Cisplatin + Herceptin (6 mg/kg) | Capecitabine + Cisplatin + Herceptin (10 mg/kg)
Serious Adverse Events (participants affected / at risk) | 35/147 | 38/147
Other Adverse Events (participants affected / at risk) | 123/147 | 122/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Cisplatin + Herceptin (6 mg/kg) (N=147) | Capecitabine + Cisplatin + Herceptin (10 mg/kg) (N=147)
Anemia (Blood and lymphatic system disorders) | 7 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Obstruction gastric (Gastrointestinal disorders) | 2 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 3
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Infective spondylitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 2 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Lymphatic duct injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Renal failure (Renal and urinary disorders) | 3 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Cisplatin + Herceptin (6 mg/kg) (N=147) | Capecitabine + Cisplatin + Herceptin (10 mg/kg) (N=147)
Anaemia (Blood and lymphatic system disorders) | 47 | 40
Leukopenia (Blood and lymphatic system disorders) | 26 | 24
Neutropenia (Blood and lymphatic system disorders) | 61 | 69
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 14
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Abdominal pain upper (Gastrointestinal disorders) | 12 | 11
Constipation (Gastrointestinal disorders) | 19 | 25
Diarrhoea (Gastrointestinal disorders) | 24 | 30
Nausea (Gastrointestinal disorders) | 55 | 55
Vomiting (Gastrointestinal disorders) | 36 | 42
Asthenia (General disorders) | 16 | 11
Fatigue (General disorders) | 25 | 23
Oedema peripheral (General disorders) | 9 | 6
Pyrexia (General disorders) | 15 | 14
Weight decreased (Investigations) | 10 | 17
Decreased appetite (Metabolism and nutrition disorders) | 32 | 27
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 8
Dizziness (Nervous system disorders) | 8 | 2
Chronic kidney disease (Renal and urinary disorders) | 7 | 13
Renal failure (Renal and urinary disorders) | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 | 20

LIMITATIONS AND CAVEATS:
Trial was stopped for futility based on pre-planned interim analysis results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.